CLINICAL TRIAL: NCT03242369
Title: Comparison of the Effectiveness of Bowel Preparations in Bowel Cleansing Before Colonoscopy - Prospective, Randomized Study
Brief Title: Comparison of the Effectiveness of Bowel Preparations Before Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military University Hospital, Prague (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Stepan Suchanek, MD., Ph.D., Head of Department of Gastrointestinal Endoscopy, Military University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 108/11-29/2017
Record Dates: First submitted 2017-07-18; First posted 2017-08-08 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal neoplasia; colonoscopy; quality of bowel cleansing; bowel preparation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PEG group (Experimental): 100 patients undergoing colonoscopy.
  Interventions: Procedure: colonoscopy
- SBS group (Experimental): 100 patients undergoing colonoscopy
  Interventions: Procedure: colonoscopy
- PEG 2L + ascorbic acid group (Experimental): 100 patients undergoing colonoscopy.
  Interventions: Procedure: colonoscopy
- PICO group (Experimental): 100 patients undergoing colonoscopy.
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: colonoscopy — 100 patients undergoing colonoscopy will be prepared with split dose (2+2l) PEG. 2 liters will be drunk during 2 hours in the evening the day before colonoscopy, the second 2l during 2 hours in the day of colonoscopy finishing the dose 4- 6 hours before colonoscopy.
  Arms: PEG group
Procedure: colonoscopy — 100 patients undergoing colonoscopy will by prepared with split dose of SS. The first bottle of SS with water (total volume 0,5l) will be drunk in the evening the day before colonoscopy during 1 hour, than another 1liter of clear fluid will be drunk. The same procedure will be repeated with the second bottle of SS finishing at least 3 hours before colonoscop
  Arms: SBS group
Procedure: colonoscopy — 100 patients undergoing colonoscopy will be prepared with split dose of PEG (1+1L) with ascorbic acid. The first 1l of solution will be drunk in the evening the day before colonoscopy, the second 1l of solution in the day of colonoscopy finishing 4-6 hours before the examination. Another 1l of clear fluid should be drunk during the cleansing process.
  Arms: PEG 2L + ascorbic acid group
Procedure: colonoscopy — 100 patients undergoing colonoscopy will be prepared with split dose (150ml +150ml) of solution of magnesium acid and sodium picosulfate. The first dose will be drunk in the evening the day before colonoscopy, then at least 1l of another clear fluid will be drunk within a few hours, the second dose will be drunk in the day of examination finishing 4-6hours before colonoscopy and then another at least 750ml clear fluid.
  Arms: PICO group

SUMMARY:
Polyethylene glycol is the gold standard of bowel preparation for colonoscopy. The most important disadvantage is high volume of this preparation. Sulphate based solution (SBS), low volume PEG + ascorbic acid and solution of magnesium citric acid and sodium picosulfate could be suitable substitution of polyethylene glycol.

DETAILED DESCRIPTION:
This study will be unicenter, randomized and single blind. It focuses on studying the effectiveness of four preparations for bowel cleansing before colonoscopy. Polyethylenglycol (PEG) will be compared as a gold standard of bowel cleansing with low volume preparations: Sulfate-based solution (SBS), low volume PEG + ascorbic acid and solution of magnesium citric-acid and sodium picosulfate. The effectiveness will be rated according to a quality of bowel preparation (Boston Bowel Preparation Scale) and detection of a colorectal neoplasia. The aim of this project is to compare the effectiveness of each four preparations.

Primary endpoint: To compare a quality of bowel preparation. Secondary endpoint: To compare a detection of colorectal neoplasia in those preparations.

Main hypothesis: PEG as a gold standard of bowel cleansing preparation is not worse than the other compared preparations.

Secondary hypothesis: PEG is not worse in detection of colorectal neoplasia than the other compared preparations.

Methods: There will be 400 patients included in the project with all indications for colonoscopy (age ≥ 18 years, no upper age limit) except the exclusion criteria. The patients will be offered to participate in the study at the Endoscopy unit when arranging the examination. In case of agreement they will sign informed consent and they will be educated about the correct process of bowel preparation. They also get all the instructions in printed version and questionnaire of preparation tolerability. The advantages for the patients in study will be earlier date of colonoscopy. On the day of colonoscopy, the patients will submit the questionnaire and undergo standard colonoscopy examination.

The quality of a bowel cleansing will be evaluated by the experienced endoscopists who will be blinded about a type of bowel preparation. The effectiveness will be assessed by the degree of bowel cleansing (Boston Bowel Preparation Scale) and ADR, aADR and number of cancers diagnosed. The GE unit staff will record all results in the on-line study database. Results will be statistically evaluated in Institute of Biostatistics and Analyses, Masaryk University, IBA MU).

ELIGIBILITY:
Inclusion Criteria:

• Individuls ≥ 18 years old undergoing colonoscopy for all indications except exclusion criteria

Exclusion Criteria:

* Active idiopathic bowel disease
* Chronic renal insufficiency
* Serious internal comorbidity
* Planned therapeutic colonoscopy
* No informed consent signed (with the study and/or with the colonoscopy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Quality of bowel cleansing according to Boston Bowel Preparation Scale (BBPS) | 1 day
  * 0-Unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared
  * 1-Portion of mucosa of the colon segment seen, but other areas of the segment are not well seen due to staining, residual stool, and/or opaque liquid
  * 2-Minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa colon segment is seen well
  * 3-Entire mucosa of colon segment seen well, with no residual staining, small fragment of stool or opaque liquid

SECONDARY OUTCOMES:
Detection of colorectal neoplasia | 1 day
  In each colonoscopy the number of colorectal neoplasia will be rated.
  Colorectal neoplasia is defined by these two types of lession:
  * advanced adenoma - 1cm size or greater or with villous component or with high grade dysplasia
  * carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Stepan Suchanek, MD., PhD., Study Director — Military Univesity Hosital Prague
Locations (1):
- Military University Hospital, Prague, Czechia